CLINICAL TRIAL: NCT03067220
Title: Can A Virtual Clinic Review Replace A Surgical Clinic Visit After Discharge?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connolly Hospital Blanchardstown (Other)
Responsible Party: Principal Investigator, Paul Healy, Surgical Registrar, Connolly Hospital Blanchardstown
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ConnollyHB
Record Dates: First submitted 2017-02-22; First posted 2017-03-01 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Outpatients General Surgery Virtual Clinic
Keywords: outpatients; general surgery; virtual clinic; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard outpatient clinic appointment (Other): Patients will be sent an appointment letter to return to a scheduled outpatient clinic for review approximately 6 weeks after their discharge from hospital
  Interventions: Other: Standard outpatient clinic appointment
- Virtual out patient clinic appointment (Experimental): Patients will be sent an appointment letter stating a specific day approximately 6 weeks after their discharge from hospital in which they will be contacted by telephone for a review by a junior doctor from the discharging team.
  Interventions: Other: Virtual outpatient clinic appointment

INTERVENTIONS:
Other: Virtual outpatient clinic appointment — Patients will be sent an appointment letter stating a specific day approximately 6 weeks after their discharge from hospital in which they will be contacted by telephone for a review by a junior doctor from the discharging team.
  Arms: Virtual out patient clinic appointment
Other: Standard outpatient clinic appointment — Patients will be sent an appointment letter to return to a scheduled outpatient clinic for review approximately 6 weeks after their discharge from hospital
  Arms: Standard outpatient clinic appointment

SUMMARY:
To assess if a virtual out patient clinic via a telephone review was an acceptable and safe alternative to a clinic attendance for a broad range of general surgical patients discharged following a hospital admission.

DETAILED DESCRIPTION:
The surgical out patients is often the first point of contact between a surgeon and patient after being referred by their general practitioner (GP). Here new patients are assessed, investigations are requested and treatment plans devised. On completion of treatment it has been common practice to review all patients post operatively (1). However the routine review of patients following low risk procedures contribute to increasing healthcare costs without necessarily a significant benefit for the patient. It may indeed be a burden on patients and families, who may miss work or college, have to travel long distances and wait for prolonged periods to be seen. There is also a financial burden associated with travel to appointments and on-site parking fees. Unnecessary appointments also contribute to increased waiting times for new referrals to be seen. This has the potential to lead to delayed diagnosis of serious conditions (2) and further increase the workload of overburdened emergency departments.

Previous studies have demonstrated a safe and acceptable alternative to traditional outpatient appointments with telephone follow up in certain paediatric and adult surgical patients (1,3,4). Improved efficiency and high levels of patient satisfaction have also been demonstrated in an Irish setting with the establishment of a virtual outpatient department (VOPD) following endoscopy (5). In an oncology setting telephone follow up has also been identified as an effective means of delivering care (6,7). In particular nurse led follow up of lung, breast and colorectal cancer patients has been associated with a high level of patient satisfaction (8).

The aim of this study was to determine whether a virtual out patient clinic via a telephone review was an acceptable and safe alternative to a clinic attendance for a broad range of general surgical patients discharged following a hospital admission.

If eligible for inclusion the patient was approached prior to discharge and the study rationale, randomisation and methods of follow up were explained. If they agreed to participate written consent was obtained and an information leaflet about the study was provided. Randomisation was performed by selecting an unmarked white envelope which contained either a coloured card indicating a telephone call follow up within 6-8 weeks or a white card indicating follow up with an outpatient appointment at 6-8 weeks.

After randomisation the patient was provided with a letter detailing their specific follow up arrangements and a contact number was provided if they had any further questions after discharge. Patients' were sent a further letter by administration staff after discharge, with the specific date of either the clinic appointment or phone follow up.

ELIGIBILITY:
Inclusion Criteria:

* Over 16 years old
* Could provide written consent
* Comprised one of four categories based on reason for admission

  * Category 1 - minor surgery
  * Category 2- elective or emergency surgery such as appendicectomy, hernia repair, thyroidectomy
  * Category 3- admitted for investigation or management of conditions such as non specific abdominal pain, head injury, cellulitis
  * Category 4- attended for surveillance endoscopy for conditions such as colonic polys or Barrett's oesophagus

Exclusion Criteria:

* Declined to participate
* Had a previous, new or suspected diagnosis of malignancy
* On-going issues requiring follow up such as wound healing problems
* Required further investigation such as endoscopy after admission with e.g. diverticulitis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the rate of complications or on going issues requiring further assessment in either group. | At each patients review appointment approximately 6 weeks after discharge.
  Any unexpected outcome reported by the patient if contacted by telephone or reported and assessed by a doctor on their review at a standard clinic appointment. This would be expected to be an issue resulting in a deviation from a normal and expected post discharge recovery.

SECONDARY OUTCOMES:
Secondary outcomes included a "did not respond" (DNR) or did not attend (DNA) rate | At each patients review appointment approximately 6 weeks after discharge.
  If an attempt to contact the patient by telephone to conduct their review appointment is unsuccessful this will be recorded as a did not respond. A DNA will be recorded if a patient fails to attend for their scheduled review appointment
The number of patients listed for further procedures, investigation or referral to other specialities based on their review. | At each patients review appointment approximately 6 weeks after discharge.
  If the patient is not discharged from follow up by the hospital service to the care of their general practitioner, these are the anticipated outcomes of the follow up review for each patient not discharged
Patient satisfaction and opinions regarding their follow up arrangements | 6-8 weeks after their review appointment
  Questionnaire that allows participants to provide free text responses about their experience.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walsh, MD MCh FCRSI, Study Chair — Department of General Surgery, Connolly Hospital and Royal College of Surgeons in Ireland
Locations (1):
- Connolly Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McVay MR, Kelley KR, Mathews DL, Jackson RJ, Kokoska ER, Smith SD. Postoperative follow-up: is a phone call enough? J Pediatr Surg. 2008 Jan;43(1):83-6. doi: 10.1016/j.jpedsurg.2007.09.025. PMID 18206461
- [Background] Allgar VL, Neal RD. Delays in the diagnosis of six cancers: analysis of data from the National Survey of NHS Patients: Cancer. Br J Cancer. 2005 Jun 6;92(11):1959-70. doi: 10.1038/sj.bjc.6602587. PMID 15870714
- [Background] Gray RT, Sut MK, Badger SA, Harvey CF. Post-operative telephone review is cost-effective and acceptable to patients. Ulster Med J. 2010 May;79(2):76-9. PMID 21116423
- [Background] Rosbe KW, Jones D, Jalisi S, Bray MA. Efficacy of postoperative follow-up telephone calls for patients who underwent adenotonsillectomy. Arch Otolaryngol Head Neck Surg. 2000 Jun;126(6):718-21; discussion 722. doi: 10.1001/archotol.126.6.718. PMID 10864107
- [Background] Ryan EM, Rogers AC, Hanly AM, McCawley N, Deasy J, McNamara DA. A virtual outpatient department provides a satisfactory patient experience following endoscopy. Int J Colorectal Dis. 2014 Mar;29(3):359-64. doi: 10.1007/s00384-013-1801-y. Epub 2013 Dec 6. PMID 24309978
- [Background] Sardell S, Sharpe G, Ashley S, Guerrero D, Brada M. Evaluation of a nurse-led telephone clinic in the follow-up of patients with malignant glioma. Clin Oncol (R Coll Radiol). 2000;12(1):36-41. doi: 10.1053/clon.2000.9108. PMID 10749018
- [Background] Booker J, Eardley A, Cowan R, Logue J, Wylie J, Caress AL. Telephone first post-intervention follow-up for men who have had radical radiotherapy to the prostate: evaluation of a novel service delivery approach. Eur J Oncol Nurs. 2004 Dec;8(4):325-33. doi: 10.1016/j.ejon.2004.01.003. PMID 15550362
- [Background] Beaver K, Williamson S, Chalmers K. Telephone follow-up after treatment for breast cancer: views and experiences of patients and specialist breast care nurses. J Clin Nurs. 2010 Oct;19(19-20):2916-24. doi: 10.1111/j.1365-2702.2010.03197.x. PMID 20649914